CLINICAL TRIAL: NCT05958810
Title: Efficacy and Safety of Artemether-lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Philippines in 2017-2018
Brief Title: TES of Artemether-lumefantrine for Pf in the Philippines in 2017-2018
Acronym: TES
Status: Completed | Type: Observational
Sponsor: Research Institute for Tropical Medicine, Philippines (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Fe Espino, Medical Specialist IV, Principal Investigator, Head of Parasitology Department, Research Institute for Tropical Medicine, Philippines
Other Study IDs: 2003-25-12_2017
Record Dates: First submitted 2023-06-30; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Malaria,Falciparum; Malaria Recrudescence
Keywords: Malaria; TES; Artemether-lumefantrine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Capillary blood (malaria blood film and filter paper)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients detected with Plasmodium falciparum (Artemether-lumefantrine): Patients with mono-infection of Plasmodium falciparum with 1,000-100,000 asexual forms per µl
  Interventions: Drug: Artemether-lumefantrine; Drug: Primaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Artemether-lumefantrine will be administered for 3 days according to body weight (Days 0 and 8 hours after, 1 and 2). Dosage depending on body weight or age if weight cannot be determined.
  Dosage: 1 tablet contains 20 mg artemether and 120 mg lumefantrine Dosage per weight: 1 tablet (5 to <16kg); 2 tablets (15 to <25kg); 3 tablets (25 to <35kg), 4 tablets for >35 kg) Dosage per age, if weight cannot be determined: 1 tablet (6 months old to 3 years old); 2 tablets (4 to 8 years old); 3 tablets (9-13 years old), 4 tablets (>13 years old)
  Other Names: Coartem
Drug: Primaquine — For Pf patients, primaquine at 0.75 mg base/kg body weight single dose will be given on Day 3 for Pf patients; For Pv patients primaquine will be withheld for 28 days and will be given after Day 28 follow-up, at 0.25 mg base/kg per day for 14 days.

SUMMARY:
The emergence and spread of drug resistance is a major obstacle to combating malaria. The World Health Organization (WHO) recommends that regular efficacy monitoring should be undertaken by all malaria endemic countries that have deployed artemisinin combination therapy (ACT), to help early detection of drug resistant strains of the parasite and contain their rapid spread. Artemether-lumefantrine (AL) has been the first-line antimalarial drug against uncomplicated Plasmodium falciparum malaria in the Philippines since 2009, with primaquine as an anti-relapse drug. The objective of this study is to assess the safety and efficacy of artemether-lumefantrine for the treatment of uncomplicated P. falciparum infections in the Philippines. The study was conducted in three (3) municipalities (Bataraza, Brooke's Point, and Rizal) of Palawan. Single-arm prospective study of a 28-day follow-up was conducted from February 2017 to December 2018 according to the revised WHO 2014 drug efficacy study protocol. Study subjects were consenting individuals seeking care at the selected Rural Health Units, who were aged >6 months old to 59 years old with confirmed uncomplicated P. falciparum infections. AL was administered for 3 days according to body weight (Days 0, 1 and 2) and primaquine 0.75 mg/kg body weight single dose was given on Day 3 following the National Treatment Guidelines.

DETAILED DESCRIPTION:
Early diagnosis and timely treatment of malaria with an effective drug is an important strategy to control malaria. However, antimalarial drug resistance is one of the major obstacles to controlling this disease. Following a widespread failure of chloroquine (CQ) and sulfadoxine-pyrimethamine (SP), most malaria-endemic countries had shifted their malaria treatment policy to artemisinin-based combination therapy (ACT). In the Philippines, AL became the first-line drug for falciparum malaria in the 2009 revised drug policy. The DOH in the past years (2002-2007) adopted the use of AL in the highly endemic areas of the country and conducted therapeutic efficacy studies (TES) in 3 sentinel sites: Kalinga-Isabela, Palawan and several Mindanao provinces, showing 97-100% efficacy. Whereas CQ+SP showed variability and declining efficacy, results ranged from 70%-95% (CARAGA region). In Sultan Kudarat province, results in 2006-2007 showed 90% efficacy of CQ+SP and 96% for AL for falciparum malaria. The last TES of AL as a first-line drug of choice for falciparum malaria was made in 2015 with 98.7% efficacy.

The results of this study will be used to assist the Department of Health of the Philippines in assessing the current national treatment guidelines for P. falciparum and updating the policy if necessary.

OBJECTIVES. The general objective of this study is to assess the therapeutic efficacy and safety of artemether-lumefantrine for treatment of chloroquine for the treatment of uncomplicated P. falciparum infections in the Philippines in 2017-2018.

The primary objectives are:

1. To measure the clinical and parasitological efficacy of artemether-lumenfantrine (AL) among patients aged between > 6 months and 59 years old suffering from uncomplicated falciparum malaria, by determining the proportion of patients with Early Treatment Failure (ETF), Late Clinical Failure (LTF), Late Parasitological Failure (LPF), or an Adequate Clinical and Parasitological Response (ACPR) as indicators of efficacy;
2. To differentiate recrudescences from new infections by the Polymerase Chain Reaction (PCR) analysis;

The secondary objectives are:

1. To evaluate the incidence of adverse events;
2. To formulate recommendations to enable the Department of Health to make informed decisions about the possible need for updating the current national antimalarial treatment guidelines.

STUDY DESIGN. The design of this surveillance study is a one-arm, prospective evaluation of the clinical and parasitological response to directly observed treatment for falciparum malaria. Individuals with uncomplicated malaria who met the study inclusion criteria were enrolled, treated on-site with AL, and monitored for a period of 28 days if they had falciparum malaria. The follow-up consisted of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. Study patients had been classified as therapeutic failures (early or late) or adequate responders based on the results of these assessments. The proportion of patients experiencing a therapeutic failure during the follow-up period had been used to estimate the efficacy of the study drug(s). Polymerase Chain Reaction (PCR) analysis will also help distinguishes between a true recrudescence due to treatment failure and episodes of re-infection.

STUDY AREA/SETTINGS. The study was conducted in the Rural Health Units (RHU) of Rizal, Bataraza and Brookes Point. Several factors influenced the selection of sites: (a) adequate numbers of patients with symptomatic, P. falciparum malaria; (b) willingness and availability of the selected healthcare facility staff to participate in the trial and to support the work with laboratory space; (c) access of patients to the health facility for weekly follow-ups; and (d) willingness of the Municipality Health Officer (MHO), the nurse and a trained Medical Technologist to take responsibility for conducting the trial, and security.

STUDY PARTICIPANTS. The population of interest consisted of patients aged between > 6 months to 59 years old diagnosed with uncomplicated falciparum malaria attending the study health clinic and having given, or whose parents or legal guardians had given informed consent for study inclusion and assent in children as appropriate.

ETHICAL CONSIDERATIONS Participants were recruited after the study received favorable approval of the protocol, participant information sheet, and written informed consent form from RITM Institutional Review Board (IRB). The study document versions given written approval by the IRB were used. The study was carried out according to the ethical guidelines in the Declaration of Helsinki (version 2008), applicable guidelines of ICH-GCP (E6); and applicable regulations of the Department of Health, Manila. The participant's written informed consent was secured before enrolment and prior to initiating procedures specific to this study. For potential participants below 18 years old, this consent was obtained from either parent or a legally accepted guardian. An independent witness was present during the process of obtaining informed consent from a participant or parents/legal guardian who was illiterate.

ELIGIBILITY:
Inclusion Criteria:

* Above 6 months old to 59 years old;
* Mono-infection with P. falciparum (1000-100 000 asexual forms per µl)
* Axillary temperature ≥37.5 °C or oral/rectal temperature of ≥38 °C;
* Ability to swallow medication;
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* Informed consent from the patient or from a parent or legal guardian in the case of children less than 18 years old;
* Informed assent from any minor participant aged 12 - 17 years;
* Consent for pregnancy testing from females of child-bearing potential and from their parent or guardian if under 18 years old.

Exclusion Criteria:

* Presence of general danger signs among children <5 years old or other signs of severe and complicated falciparum malaria according to current WHO definitions
* Mixed Plasmodium species;
* Presence of severe malnutrition
* Presence of febrile conditions due to diseases other than malaria (measles, acute lower tract respiratory infection, severe diarrhea with dehydration, etc.), or other known underlying chronic or severe diseases (e.g. cardiac, renal, hepatic diseases, HIV/AIDS)
* History of hypersensitivity reactions to any of the drug(s) being tested or used as alternative treatment.

Ages: 6 Months to 59 Years | Sex: All
Age Groups: Child, Adult
Study Population: The population of interest consists of patients aged between > 6 months to 59 years old diagnosed with uncomplicated falciparum malaria attending the study health clinic, and having given, or whose parents or legal guardians have given informed consent for study inclusion and assent in children as appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Early Treatment Failure (ETF) | Day 1-3
  The number of patients with the following criteria based on microscopy results without PCR:
  * Development of danger signs or severe malaria on day 1, day 2, or day 3 in the presence of parasitemia;
  * Parasitaemia on day 2 higher than day 0 count irrespective of axillary temperature;
  * Parasitaemia on day 3 with axillary temperature ≥37.5 ºC;
  * Parasitaemia on day 3 ≥25% of count on day 0.
Late Clinical Failure (LCF) | Day 4-28
  The number of patients with the following criteria based on microscopy results without PCR:
  * Development of danger signs or severe malaria on any day from day 4 to day 28 in the presence of parasitemia, without previously meeting any of the criteria of Early Treatment Failure;
  * Presence of parasitemia and axillary temperature ≥37.5 ºC (or history of fever in low/moderate transmission areas) on any day from day 4 to day 28, without previously meeting any of the criteria of Early Treatment Failure.
Number of Patients with Late Parasitological Failure (LPF) | Day 7-28
  The number of patients with the presence of parasitemia on any day from day 7 to day 28 and axillary temperature <37.5 ºC, without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure.
Number of Patients with Adequate Clinical and Parasitological Response (ACPR) | Day 0-28
  The number of patients with absence of parasitemia on day 28 irrespective of axillary temperature without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure or Late Parasitological Failure.

CONTACTS AND LOCATIONS:
Overall Officials: Fe Esperanza Caridad J Espino, MD, PhD, Principal Investigator — Research Institute for Tropical Medicine

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with Data Transfer Agreement and IRB Approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data information will be provided upon request
Access Criteria: Data Transfer

REFERENCES:
- [Background] Council for International Organizations of Medical Sciences. International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics. 2002 Oct;(182):17-23. PMID 14983848
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05958810/Prot_SAP_000.pdf